CLINICAL TRIAL: NCT02496559
Title: Children With Fever and Respiratory Symptoms at Out-of-hours Services in Norway
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lower prevalence than expected and the inclusion was difficult.
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NKLM 2012/1471 RV
Record Dates: First submitted 2015-06-25; First posted 2015-07-14 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Children
Keywords: C-reactive Protein; Primary Health Care; Child Welfare; After-Hours Care; Anti-Bacterial Agents; Drug Prescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-consultation CRP (Active Comparator): Every third child included get a CRP-test before the consultation and the doctor have the answer at start of consultation
  Interventions: Procedure: Pre-consultation CRP
- CRP requested (No Intervention): No intervention, the consultation with children as normal, the CRP is used at doctors request.

INTERVENTIONS:
Procedure: Pre-consultation CRP — Use of CRP test on all children with fever before the consultation (intervention) compared to where the doctor requests a CRP test (no intervention)
  Arms: Pre-consultation CRP

SUMMARY:
Viral self-limiting infections in respiratory organs among children are common in primary care. Serious infections have low prevalence and are challenging to distinguish from self-limiting infections.

Prescription of antibiotics in primary care is still high but stable since 2009 in Norway, and 90% of all antibiotics are prescribed in primary care.

C-reactive protein (CRP) has been especially popular in Norway for point-of-care testing in primary care, but its role in ruling-out serious infections and the cut-off value for prescribing antibiotics has been discussed a lot.

The aim of this study is to identify if pretesting with CRP of all children 0-6 year with fever or respiratory symptoms at Out-of-Hours Services will affect the prescription of antibiotics and the referral to hospital for children.

DETAILED DESCRIPTION:
Design: A randomized controlled observational study including children 0-6 year with fever and/or respiratory symptoms at 4 different Out-of-hour Services and at 1 Emergency Children Department Clinic at a hospital (open clinic). The data consist of clinical data and anamnestic information from a nurse at OOH-service collected before the consultation, the doctor's journal and a questionnaire to parents before the consultation and 1 week after the consultation.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-6 years with fever and/or respiratory symptoms

Exclusion Criteria:

* Children older than 6 years with other conditions

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 401 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescription rate | 24 hours
  Number of participants prescribed antibiotics

SECONDARY OUTCOMES:
Hospitalization rate | 24 hours
  Number of participants referred to hospital
Rate of side-effects of antibiotics | 7 days
  Number of participants with side-effects of antibiotics prescribed at Out-of-hours Service
Duration of illness | 7 days
  Number of days with fever and respiratory symptoms after the consultation at the Out-of-hours Service.

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Hunskår, Prof. dr.med, Study Director — NORCE Norwegian Research Centre AS

REFERENCES:
- [Background] Brent AJ, Lakhanpaul M, Thompson M, Collier J, Ray S, Ninis N, Levin M, MacFaul R. Risk score to stratify children with suspected serious bacterial infection: observational cohort study. Arch Dis Child. 2011 Apr;96(4):361-7. doi: 10.1136/adc.2010.183111. Epub 2011 Jan 24. PMID 21266341
- [Background] Van den Bruel A, Thompson MJ, Haj-Hassan T, Stevens R, Moll H, Lakhanpaul M, Mant D. Diagnostic value of laboratory tests in identifying serious infections in febrile children: systematic review. BMJ. 2011 Jun 8;342:d3082. doi: 10.1136/bmj.d3082. PMID 21653621
- [Background] Nordlie AL, Andersen BM. [Changes in antibiotic consumption among day-care children in Oslo]. Tidsskr Nor Laegeforen. 2007 Nov 15;127(22):2924-6. Norwegian. PMID 18026237
- [Result] Rebnord IK, Sandvik H, Hunskaar S. Use of laboratory tests in out-of-hours services in Norway. Scand J Prim Health Care. 2012 Jun;30(2):76-80. doi: 10.3109/02813432.2012.684208. PMID 22643151
- [Result] Magnus MC, Vestrheim DF, Nystad W, Haberg SE, Stigum H, London SJ, Bergsaker MA, Caugant DA, Aaberge IS, Nafstad P. Decline in early childhood respiratory tract infections in the Norwegian mother and child cohort study after introduction of pneumococcal conjugate vaccination. Pediatr Infect Dis J. 2012 Sep;31(9):951-5. doi: 10.1097/INF.0b013e31825d2f76. PMID 22627867
- [Derived] Alvsaker LKT, Stensen MF, Mjelle AB, Hunskaar S, Rebnord IK. Outcomes of antibiotic treatment for respiratory infections in children an observational study in primary care. Scand J Prim Health Care. 2024 Jun;42(2):237-245. doi: 10.1080/02813432.2024.2305929. Epub 2024 Jan 24. PMID 38265029
- [Derived] Rebnord IK, Sandvik H, Mjelle AB, Hunskaar S. Factors predicting antibiotic prescription and referral to hospital for children with respiratory symptoms: secondary analysis of a randomised controlled study at out-of-hours services in primary care. BMJ Open. 2017 Jan 17;7(1):e012992. doi: 10.1136/bmjopen-2016-012992. PMID 28096254
- [Derived] Rebnord IK, Sandvik H, Mjelle AB, Hunskaar S. Out-of-hours antibiotic prescription after screening with C reactive protein: a randomised controlled study. BMJ Open. 2016 May 12;6(5):e011231. doi: 10.1136/bmjopen-2016-011231. PMID 27173814
- See also: Project web page — http://uni.no/en/uni-health/national-centre-for-emergency-primary-health-care/diagnostic-equipment-at-norwegian-out-of-hours-services/